CLINICAL TRIAL: NCT02159222
Title: Sepsis Trial of Early Physical Therapy Outside the ICU: A Pilot Feasibility Study
Brief Title: Sepsis Trial of Early Physical Therapy Outside the ICU
Acronym: STEP TO IT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey Rohde, Associate Professor of Internal Medicine, Medical School, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UM-HUM00073474
Record Dates: First submitted 2014-05-22; First posted 2014-06-09 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Additional physical therapy (Experimental)
  Interventions: Procedure: Additional physical therapy

INTERVENTIONS:
Procedure: Additional physical therapy

SUMMARY:
The purpose of this study is to determine whether an additional physical therapy program can improve the mobility and functional outcomes of patients diagnosed with severe sepsis (an illness in which the body has a severe response to bacteria or other germs and develops worsened function of a major organ such as the kidneys, heart, or lungs).

DETAILED DESCRIPTION:
Patients who are admitted to the hospitalist service at the University of Michigan Hospital will be screened for the presence of severe sepsis. Those who are deemed eligible and provide consent will be enrolled. Study patients will receive additional physical therapy according to a protocol developed for this study in addition to the usual care recommended by their regular treating physician. Additional treatments will be individualized based on enrolled patients' baseline physical function and progress and may include standing, stretching, transferring, and walking - either with assistance or independently. Treating therapists have been trained in the use of the protocol and individualization to maintain the highest standard of patient safety. Patients will be contacted 30 days after discharge to answer questions about their health and ability to perform routine tasks at home.

ELIGIBILITY:
Inclusion Criteria:

* Any English-speaking patient over the age of 18 who is currently admitted to a general care floor under the care of the Medicine Faculty Hospitalist Service at the University of Michigan Health System and has severe sepsis is eligible to take part in this study.

Exclusion Criteria:

* Subjects must be deemed by the study team to give informed consent by being able to state the basic purpose of the study. Consent by a legally authorized representative (LAR) will not be sought.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-04; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline ambulation | At day 0 (baseline enrollment) and for the duration of the participants' hospitalization, a predicted average length of stay of 5 days.
  Participants will be followed for the duration of their hospitalization, a predicted average length of stay of 5 days. This outcome will be assessed at baseline and at each study protocol physical therapy session during the index hospitalization.

SECONDARY OUTCOMES:
Change in Activities of Daily Living (ADLs) and Instrumental Activities of Daily Living (iADLs) | At day 0 (baseline enrollment) and day 35 (assessed at 30 days post discharge; predicted average length of stay is 5 days)
  Baseline ADLs will be assessed using chart review. 30 day follow-up ADL and iADL function will be assessed using a telephone survey
Discharge location | At day 5 (assessed at discharge; predicted average length of stay is 5 days)
  The location of discharge (home, subacute rehabilitation facility, skilled nursing facility) will be assessed at discharge for all patients enrolled in the study.
ICU Transfer Rate | Participants will be followed for the duration of their hospitalization, an average length of stay of 5 days.
  The rate at which patients require transfer to the ICU will be assessed.
Length of stay | Participants will be followed for the duration of their hospitalization, a predicted average length of stay of 5 days.
  The length of stay will be recorded for patients enrolled in the trial.
Employment status | At day 35 (assessed at 30 days post discharge; predicted average length of stay is 5 days).
  For patients employed for pay prior to the index admission, employment status will be assessed by telephone survey 30 days post-discharge.
Post-hospitalization physical function | At day 35 (assessed at 30 days post discharge; predicted average length of stay is 5 days).
  Patients' physical function will be assessed 30 days after discharge using the SF-10 instrument.

OTHER OUTCOMES:
Readmission | At day 35 (assessed at 30 days post discharge; predicted average length of stay is 5 days).
In-Hospital Mortality | Participants will be followed for the duration of their hospitalization, a predicted average length of stay of 5 days
Falls | Participants will be followed for the duration of their hospitalization, a predicted average length of stay of 5 days.
Arrhythmia | During each study protocol physical therapy session while hospitalized
  Clinically significant arrhythmias occurring during therapy sessions will be documented and recorded as a safety outcome.
Pressure ulcers | Participants will be followed for the duration of their hospitalization, a predicted average length of stay of 5 days.
  The presence and severity of pressure ulcers will be recorded.
Cognitive function | At day 35 (assessed at 30 days post discharge; predicted average length of stay is 5 days).
  Enrolled patients' cognitive function will be assessed using the TICS-m instrument
Depression | At day 35 (assessed at 30 days post discharge; predicted average length of stay is 5 days).
  Patients will be screened for depression using the PHQ-2 instrument as part of the follow-up telephone survey.
30-Day Post-Hospitalization Mortality | At day 35 (assessed at 30 days post discharge; predicted average length of stay is 5 days).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Odden, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States